CLINICAL TRIAL: NCT02790086
Title: Prevalence Survey in France of Unintentional Perioperative Hypothermia and Its Impact on Two Outcomes: Blood Loss, Myocardial Injury After Non Cardiac Surgery
Brief Title: Prevalence Survey in France of Unintentional Perioperative Hypothermia and Its Impact on Two Outcomes
Acronym: HYPOTHERMIE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Société Française d'Anesthésie et de Réanimation (Other)
Responsible Party: Sponsor
Other Study IDs: 13-HYPOTHERMIE
Record Dates: First submitted 2016-05-04; First posted 2016-06-03 (Estimated); Last update posted 2016-06-03 (Estimated); Status verified 2016-05

CONDITIONS: Hypothermia, Perioperative
Keywords: hypothermia; prevalence; perioperative; anemia; myocardial injury; troponin T; noncardiac surgery
MeSH Terms: conditions — Hypothermia; Anemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 2 tubes of 5 ml of blood
Oversight: Data Monitoring Committee: No

SUMMARY:
The primary objectives of the study are

* to perform a survey on the clinical management of unintentional hypothermia during surgery in France.
* to assess the impact of perioperative hypothermia on anemia and myocardial injury.

DETAILED DESCRIPTION:
100 investigation centers in metropolitan France will participate in the study, targeting 2000 included patients (20 surgical interventions in each center). The duration of inclusion in each center should last at most 2 weeks.

The selected surgical interventions will be those performed with a high frequency, practiced in all types of hospitals (public, private, university hospital or not), and requiring anesthesia of at leat 30 minutes (general, epidural or intrathecal anesthesia).

ELIGIBILITY:
Inclusion criteria:

* Non-ambulatory surgery.
* Duration of anesthesia > 30 minutes.
* Type of surgery: urology, gynecological, gastrointestinal, vascular and orthopedics surgery.
* Type of anesthesia: general, intrathecal or epidural anesthesia.
* patient ≥ 45 years.
* No opposition of patient to participate in the study.

Exclusion criteria:

* Emergency surgery.
* Cardiac surgery, proctology surgery or thoracic surgery.
* Digestive endoscopy or surgical radiology.
* Septic surgery.
* Patient with at least one organ failure.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing surgical intervention, requiring 2 days of hospitalization
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2014-10; Primary Completion 2016-07 (Estimated); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
Core temperature | up to 24 hours
  The temperature will be measured with the same type of thermometer in all investigator sites: SpotOn™ (3M France).
blood loss | up to 24 hours
  Blood loss will be assessed by haemoglobin variation between preoperative and the first post-operative day.
myocardial injury | up to 48 hours
  Troponin T will be measured after the surgical intervention (at least 6 hours after the end of the surgery) and on the second postoperative day (when the patient remains hospitalized).

CONTACTS AND LOCATIONS:
Overall Officials: Pascal ALFONSI, MD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Service d'Anesthésie-Réanimation Chirurgicale, Hôpital Cochin, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No